CLINICAL TRIAL: NCT06090214
Title: Circulating Tumor Cells for the Diagnosis of Intestinal-type Adenocarcinoma of the Ethmoid : a Pilot Study
Brief Title: Liquid Biopsy for the Diagnosis of Intestinal-type Adenocarcinoma of the Ethmoid (BLADE)
Acronym: BLADE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: GEFLUC Occitanie (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL22_0025
Record Dates: First submitted 2023-10-05; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Ethmoid Sinus Tumor; Adenocarcinoma; Circulating Tumor Cell
MeSH Terms: conditions — Adenocarcinoma; Neoplastic Cells, Circulating | interventions — Liquid Biopsy

STUDY DESIGN:
Intervention Model Description: The subjects will be included in the 3 following groups :
  Group 1 : Patients: n=14 Group 2 : Controls, exposed to the same occupational risks n=14 Group 3 : unexposed controls n=14
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cases: adenocarcinoma of the ethmoid Group1 (Experimental): Liquid biopsy at the inclusion (V0), d8-d10 (V1) and m2-m3 (V2) of postoperative follow-up.
  Interventions: Diagnostic Test: Liquid biopsy
- Age-matched controls Group 2 (Active Comparator): Liquid biopsy at the inclusion (V0) only
  Interventions: Diagnostic Test: Liquid biopsy
- Exposition-matched controls Group 3 (Active Comparator): Liquid biopsy at the inclusion (V0) only
  Interventions: Diagnostic Test: Liquid biopsy

INTERVENTIONS:
Diagnostic Test: Liquid biopsy — For cases: 60 mL blood sample (40 ml for CellSave analysis and 20ml for collection) at visit1 then 20 ml for CellSave analysis at visit2 and visit3 For controls: 40 ml (20ml for CellSave analysis and 20ml for collection) at visit1

SUMMARY:
The role of this transversal study is to assess the specificity and sensitivity of liquid biopsy to detect circulating cells tumor of adenocarcinoma of the ethmoid.

Blood sample of participants will be collected at the moment of the surgical procedure or recurrence diagnosis; immediately after surgery; at day 8-10; at month 2-3 of postoperative follow-up.

Two comparison groups will be studied: one age and gender-matched group and one professional exposure-matched group to assess the sensitivity and specificity of liquid biopsy

ELIGIBILITY:
Inclusion Criteria:

* Case group: diagnosis of adenocarcinoma of the ethmoid on biopsy or imaging recurence; age>/= 18 years; patient consent ;
* Age and gender-matched control group: consulting patient in otolaryngology head and neck surgery department without adenocarcinoma of the ethmoid; no personal history of cancer; no familial history of colorectal adenocarcinoma;
* Exposition control group: Professional exposition to wood dust, leaver or nickel for at least 12 months; consulting patient in otolaryngology head and neck surgery department without adenocarcinoma of the ethmoid; no personal history of cancer; no familial history of colorectal adenocarcinoma;

Exclusion Criteria:

* patient presenting with another malignant tumor
* deprivation of liberty
* patient under guardianship
* Other cancer diagnosed or under treatment
* Recurrent patient previously included in the study
* Refusal to accept the monitoring described and/or to provide the information required for the study
* No affiliation or non-beneficiary of a Social Security system;
* Pregnant or breast-feeding women in accordance with article L1121-5 of the Public Health Code (CSP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of circulating tumor cell | Day0, Day 7 to 10, VMonth 3 for patients ; Day 0 for controls
  Presence of at least 1 circulating tumor cell in the liquid biopsies

SECONDARY OUTCOMES:
Number of postoperative circulating tumor cell release | At the surgery
  Change of number circulating tumor cells detection in the liquid biopsy after surgery
Tumor Node Metastasis (TNM) classification | Day 0
  Description of TNM classification
Tumor diagnosis | Day 0
  Primary diagnosis or tumor recurrence
Histological subtype | Day 0
  Description of histological subtype
Presence of Circulating Tumor Cells (CTCs) in at least one of the patient's peripheral samples | at the surgery, day7, month3
  Presence of CTCs in at least one of the patient's peripheral samples
Estimated tumour volume | Day 0
  Estimated tumour volume by imaging
Location of tumour site | Day 0
  Location of tumour site (clinical, during surgery) to be plotted on a diagram